CLINICAL TRIAL: NCT00835341
Title: A Cohort Study on Prediction of Malignant Transformation of Oral Epithelial Dysplasia by p16 Methylation
Brief Title: Methylation of p16 CpG Island And Malignant Transformation of Oral Epithelial Dysplasia
Status: Completed | Type: Observational
Sponsor: Peking University (Other)
Responsible Party: Principal Investigator, Dajun Deng, Professor and Department Director, Peking University
Other Study IDs: CPDHS-434
Record Dates: First submitted 2009-02-02; First posted 2009-02-03 (Estimated); Results first posted 2010-02-23 (Estimated); Last update posted 2015-06-01 (Estimated); Status verified 2015-05

CONDITIONS: Oral Epithelial Dysplasia, Mild or Moderate Grade
Keywords: oral epithelial dysplasia; p16 methylation; prognosis; malignant transformation; oral squamous cell carcinoma
MeSH Terms: conditions — Lymphoma, Follicular; Squamous Cell Carcinoma of Head and Neck

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tissue specimen are collected from outpatients and inpatients with oral leukoplakia by biopsy or surgical resection, fixed in neutral buffered formalin, and embedded in paraffin. Genomic DNA is extracted from tissue sections.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- p16-methylated: patients with mild or moderate oral epithelial dysplasia containing methylated p16 CpG island.
- p16-unmethylated: patients with mild or moderate oral epithelial dysplasia NOT containing methylated p16 CpG island.

SUMMARY:
Oral epithelial dysplasia (OED) is one of the common precancerous lesions among Chinese adults. Biomarker is not available for detection of malignant potential of OED till now. p16 is an important tumor suppressor gene, which is inactivated frequently by methylation of CpG island in early stage of carcinogenesis. The present cohort study is to investigate whether p16 methylation is correlated with malignant transformation of OED.

DETAILED DESCRIPTION:
* Background: Identification of malignant potential of oral epithelial dysplasia (OED) is virtually impossible on histopathological grounds alone. Inactivation of p16 gene by CpG methylation is an early frequent event during oral carcinogenesis. To investigate the predictive value of p16 methylation on malignant potential in OED, we carried out the prospective cohort study.
* Methods: 101 patients with histologically confirmed mild or moderate OED were included in the present study. Baseline information of p16 methylation status of the OED lesions from 93 cases was obtained by methylation-specific PCR. Progression of the OEDs lesions was examined in 78 cases histologically during the 45.8 months double-blind followup survey (78/93). The association between p16 methylation and progression of OED was analyzed with SPSS13.0 software. All P-values were two-sided.

ELIGIBILITY:
Inclusion Criteria:

* histological diagnosis of mild or moderate grade OED; and
* enough amount of tissue sample from OED lesion for genomic DNA extraction; and
* available of methylation status of p16 CpG island in the extracted DNA sample.

Exclusion Criteria:

* histological diagnosis of severe grade OED or malignant disease; or
* amount of tissue sample is not enough for preparation of genomic DNA (20ng); or
* quality of the prepared DNA is not good enough for detection of p16 methylation; or
* OED treatment history by LASER, radiotherapy, or chemotherapy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 101 patients with mild or moderate OED were selected from cases with oral leukoplakia, lichen planus, or chronic discoid erythematosus at Peking University School of Stomatology between 1995 and 2005. All of the patients with OED had been diagnosed pathologically by at least two senior pathologists using the criteria from '2005 WHO Classification System' (Gale et al, 2005). All cases involved primary lesions without any LASER, radiation therapy or chemotherapy. p16 methylation status of OED samples was analyzed with methylation-specific PCR combined with denatured high performance liquid chromatography (Sun et al, 2004). 93 eligible cases with p16-methylated or p16-unmethylated OED were enrolled into the cohort study.
Sampling Method: Probability Sample
Enrollment: 93 (Actual)
Dates: Start 2005-03; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dajun Deng, MD, Study Director — Beijing Cancer Hospital/ Institue, Peking University School of Oncology; Hongwei Liu, MD, PhD, Principal Investigator — Peking University School of Stomatology
Locations (1):
- Department of Oral Medicine, Peking University School and Hospital of Stomatology, Beijing, China

REFERENCES:
- [Background] Gale N, Westra W, Pilch BZ, et al. Epithelial precursors lesions. In: Barnes L, Eveson JW, Reichart P, et al. eds. World Health Organization Classification of Tumors: Pathology and Genetics of Head and Neck Tumors. IARC Press, Lyon (France); 2005: 177-179.
- [Background] Sun Y, Deng D, You WC, Bai H, Zhang L, Zhou J, Shen L, Ma JL, Xie YQ, Li JY. Methylation of p16 CpG islands associated with malignant transformation of gastric dysplasia in a population-based study. Clin Cancer Res. 2004 Aug 1;10(15):5087-93. doi: 10.1158/1078-0432.CCR-03-0622. PMID 15297411
- [Result] Cao J, Zhou J, Gao Y, Gu L, Meng H, Liu H, Deng D. Methylation of p16 CpG island associated with malignant progression of oral epithelial dysplasia: a prospective cohort study. Clin Cancer Res. 2009 Aug 15;15(16):5178-83. doi: 10.1158/1078-0432.CCR-09-0580. Epub 2009 Aug 11. PMID 19671846
- See also: Beijing Cancer Hospital/ Institute, Peking University School of Oncology — http://www.bjcancer.org
- See also: Peking University School of Stomatology — http://ss.bjmu.edu.cn

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | p16-methylated | p16-unmethylated
Started | 35 | 58
Completed | 32 | 46
Not Completed | 3 | 12
Not completed — Lost to Follow-up | 3 | 12

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | p16-methylated | p16-unmethylated | Total
Number analyzed (Participants) | 35 | 58 | 93
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 23 | 39 | 62
  >=65 years | 12 | 19 | 31
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.5 (12.0) | 57.9 (11.0) | 57.7 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 36 | 57
  Male | 14 | 22 | 36
Region of Enrollment [Number; unit: participants]
  China | 35 | 58 | 93

OUTCOME MEASURES:

1. Primary Outcome: The Number of Participants With Both Clinical and Histological Evidence of Malignant Transformation of Oral Epithelial Dysplasia
Description: The follow-up examination was carried out with a 3-month interval. Re-biopsy was done as clinically indicated, e.g. the lesion recurs or has tendency for malignant development. Pathologic diagnosis was made by at least two pathologists without the knowledge of baseline p16 methylation, based on the World Health Organization's criteria, at Peking University School of Stomatology. The number of participants with malignant transformation of oral dysplasia was calculated based on the number of participants with oral dysplasia progressed to carcinoma by the end of the trial in each cohorts.
Time Frame: from 3 months to 124 months
Measure: Number; unit: participants
Arm/Group | p16-methylated | p16-unmethylated
Number analyzed (Participants) | 35 | 58
participants | 32 | 46

2. Secondary Outcome: Cancer-free Survival Time for Patients With Oral Epithelial Dysplasia
Time Frame: from 3 months to 124 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Description: All participants only got regular examinations during the followup period. No extra treatment was administrated.
Arm/Group | p16-methylated | p16-unmethylated
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/58
Other Adverse Events (participants affected / at risk) | 0/35 | 0/58

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No